CLINICAL TRIAL: NCT04803071
Title: Omega-3 Unsaturated Fatty Acid Improves Cognitive Function in Patients With Depression: a 12 Week Randomized, Double-blind, Placebo-controlled Study
Brief Title: Omega-3 Unsaturated Fatty Acid Improves Cognitive Function in Patients With Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Psychiatric Hospital (Other Government)
Responsible Party: Principal Investigator, Kangguang Lin, Dr., Guangzhou Psychiatric Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: guangzhou brain ω-3
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Cognitive Impairment; Depression
MeSH Terms: conditions — Cognitive Dysfunction; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Adjuvant therapy trial group (Experimental): N-3pufas improved cognitive formula adjuvant therapy intervention group
  Interventions: Dietary Supplement: Experimental group of n-pufas improving cognitive formula
- Adjuvant treatment control group (Active Comparator): General fish oil formula product adjuvant treatment control group
  Interventions: Dietary Supplement: General fish oil formula product adjuvant treatment control group
- Placebo assisted treatment control group (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo assisted treatment group
- Healthy group (No Intervention)

INTERVENTIONS:
Dietary Supplement: Experimental group of n-pufas improving cognitive formula — Three times a day, one capsule of n-3pufas improvement cognitive formula capsule (once in the morning, in the evening) and routine treatment for depression, lasting for 12 weeks
  Arms: Adjuvant therapy trial group
Dietary Supplement: General fish oil formula product adjuvant treatment control group — The control group: 1 capsule of general fish oil formula (once in the morning, in the evening) three times a day, plus routine treatment for depression, lasting for 12 weeks
  Arms: Adjuvant treatment control group
Dietary Supplement: Placebo assisted treatment group — Three times a day, one capsule of placebo adjuvant therapy (once in the morning, one in the evening) and conventional treatment of depression for 12 weeks
  Arms: Placebo assisted treatment control group

SUMMARY:
The aim of this study was to evaluate the effect of n-3pufas on cognitive function in patients with depression

DETAILED DESCRIPTION:
Depression is often accompanied by cognitive impairment. At present, there is no effective drug to improve the cognitive impairment in patients with depression, and the social function and quality of life of patients are affected in varying degrees. N-3 polyunsaturated fatty acids (n-3pufas) are food products with high safety and few adverse reactions. Previous clinical trials have also suggested that n-3pufas may help to improve cognitive impairment in patients with depression, but the reported results are different. We have developed a new generation of n-3pufas optimal proportion combination products and found good cognitive improvement effect in animal models of depression. Therefore, this clinical research project will screen out the depressive patients with cognitive impairment through the cognitive function battery test (MCCB) tool for schizophrenia. On the basis of routine treatment of depression, these patients will be added with the cognitive improvement formula n-3pufas capsule developed by us to explore the effect of n-3pufas formula on cognitive impairment of depression.

ELIGIBILITY:
Inclusion Criteria:① the patients met the diagnostic criteria of dsm-5 major depressive disorder; ② aged 18-55 years; ③ Hamilton Depression Scale score of 24 items ≥ 20 points; YMRS score < 6 points; ④ the score of wms-ii spatial span (assessment of working memory) in MCCB tool was less than or equal to its mean half standard deviation; ⑤ antidepressant types had not been adjusted in recent 2 weeks; 6) right handedness; 7) primary school had no change in the types of antidepressants The patients or their family members are willing to participate in the study and sign the informed consent.

Exclusion Criteria:① Merge with any other mental disorder; ② Patients with history of brain organic disease or traumatic brain injury and physical diseases; ③ abusers of drugs, alcohol or other psychoactive substances; ④ pregnant, lactating women and postpartum women; ⑤ refractory depression; ⑥ severe suicide risk (c-ssrs assessment); ⑦ MECT treatment in recent three months; ③ continuous use of diazepam drugs in recent three months; Ⅸ long-term use of npufas in recent three months; ⑩ Long term use of anti-inflammatory drugs in the past three months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 288 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
General information | At baseline
  Including gender, age, nationality, marriage, occupation, education level, education years, physical history, drug allergy history, tobacco and alcohol use.
Clinical data | At baseline
  Including the age of the first onset, the total course of disease, the course of the disease, the number of attacks, past medical history, family history, suicide and self injury.
Cognitive function assessment | At baseline, at the end of the 4th, 8th and 12th week
  Six cognitive dimensions, including processing speed, attention, working memory, language learning and memory, visual learning and memory, and executive function, were assessed by using standardized set of computer cognitive test (MCCB) based on MCCB, together with TONI-3 and tower of London (tower of London).

CONTACTS AND LOCATIONS:
Overall Officials: kangguang Lin, PHD,MD, Principal Investigator — Guangzhou Psychiatric Hospital
Locations (1):
- Guangzhou Brain Hospital (Guangzhou Huiai Hospital), Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No